CLINICAL TRIAL: NCT06409377
Title: Effect of Dexmedetomidine on Improving Intubating Conditions Without the Use of Muscle Relaxant
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Theodor Bilharz Research Institute (Other)
Responsible Party: Principal Investigator, Moshira sayed mohamed, Assistant lecturer, Theodor Bilharz Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: PT (822)
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Intubation; Muscle Relaxation; Dexmedetomidine
Keywords: Dexmedetomidine; Intubating conditions; No muscle relaxant
MeSH Terms: interventions — Dexmedetomidine; Injections; Fentanyl; Atracurium

STUDY DESIGN:
Intervention Model Description: Patients was allocated according to the randomly generated numbers into 2 groups; 37 patients in each group. The Dexmedetomidine Group (D): Patients received dexmedetomidine (1.5 μg/kg), propofol (2mg/kg), and fentanyl (1 μg/kg). The Control Group (C): Patients received propofol (2 mg/kg), fentanyl (1 μg/kg), and atracurium (0.5 mg/kg).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: 74 Adults were enrolled in the study and randomized using computer generated random numbers and divided into two groups. For the purpose of double blinding, two investigators participated in this study; an anesthesiologist who was not participating in the study prepared the study drug infusions and was responsible for drug administration. Another anesthesiologist who was unaware of group's allocation was responsible for the intubation and data collection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Dexmedetomidine Group (D) (Experimental): Patients received dexmedetomidine (1.5 μg/kg), propofol (2mg/kg), and fentanyl (1 μg/kg).
  Interventions: Drug: Precedex 200 MCG in 2 ML Injection
- The Control Group (C) (Placebo Comparator): Patients received normal saline of volume over 10 minutes.
  Interventions: Other: C group:

INTERVENTIONS:
Drug: Precedex 200 MCG in 2 ML Injection — Patients received dexmedetomidine (1.5 μg/kg) as single injection over 10 minutes.
  Other Names: C group: Patients received propofol (2 mg/kg), fentanyl (1 μg/kg), and atracurium (0.5 mg/kg).
  Arms: The Dexmedetomidine Group (D)
Other: C group: — Patients received propofol (2 mg/kg), fentanyl (1 μg/kg), and atracurium (0.5 mg/kg).
  Arms: The Control Group (C)

SUMMARY:
Tracheal intubation is usually facilitated by the administration of anesthetic drugs including a muscle relaxant. Over the past few years, several factors have led researchers to consider omitting neuromuscular blocking agents for tracheal intubation. (1, 2) Despite the frequent use of NMBAs in clinical practice, side effects associated with NMBA use can be particularly concerning such as anaphylaxis, cardiovascular effects related to histamine release or sympathomimetic properties, Bronchospasm, and prolonged paralysis. (3) Therefore, many studies (4, 5) focused on the possibility of performing tracheal intubation without the use of neuromuscular blocking agents. The challenge was to find the correct choice and dose of induction agent, opioid, or adjuvant drug to produce adequate intubating conditions without cardiovascular side effects. Dexmedetomidine is a potent and highly selective alpha-2 receptor agonist with sympatholytic, sedative, amnestic, and analgesic properties. It inhibits sympathetic activity thus terminating the pain signals and thereby blunts the pressor response associated with laryngoscopy and endotracheal intubation.

DETAILED DESCRIPTION:
Methods: the study is designed to be prospective randomized double blinded study. 74 ASA I, II patients will be divided into 2 groups group D and group C, 37 patients in each group. Group D will receive single dose of dexmedetomidine 1.5 mcg /kg in 50 ml normal saline over 10 min IV infusion and Group C will receive 50 ml normal saline over 10 min IV infusion. Intravenous induction of anesthesia will be done using propofol (2 mg/Kg), fentanyl (1 mcg/Kg) and atracurium (0.5 mg/Kg) in the control group versus propofol (2 mg/Kg), fentanyl (1 mg/kg) and normal saline in the dexmedetomidine group. After 2 minutes of mask ventilation with 2% sevoflurane, endotracheal intubation (ETI) with 7.5mm endotracheal tube for male patients and a 7mm endotracheal tube for female patients will be performed by an experienced anesthiolgist Base line readings including heart rate (HR), systolic blood pressure (SBP), diastolic blood pressure (DBP),) will be recorded and continuous measurements will be recorded till 5 minutes after intubation. Scoring of Intubation Conditions as follows: Intubation conditions will be evaluated using a scoring system, which includes 5 factors:

score 1 2 3 4 Laryngoscope: Easy Fair Difficult Impossible Vocal cords: Open Moving Closing Closed Coughing: None Slight Moderate Severe Jaw Relaxation: Complete Slight Stiff Rigid Limb movement: None Slight Moderate Severe

The score was interpreted into 3 categories: excellent, acceptable and poor conditions:

* Excellent conditions: received a score of 1 for all the 5 factors.
* Acceptable conditions: received a score of 2 for any of the 5 factors.
* Poor conditions received a score >2 for any of the 5 factors. Both excellent and acceptable conditions was defined as successful intubations. Poor conditions was defined as failed intubations.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I, II.
* Age 18- 60 years old of both sexes.
* Mallampati I, II
* Patients undergoing elective surgery under general anesthesia and tracheal intubation.

Exclusion Criteria:

* Age < 18 years and ≥ 60 years
* Pregnancy
* Emergency surgery or full stomach
* Mallampati III , IV
* Renal or Hepatic patients
* Patients with any cardiac condition
* Patients with suspected difficult airway; e.g., high neck circumference, high body mass index (≥30 kg/m2), airway masses, mouth scars, neck scars, limited neck extension or history of snoring.
* Any patient on regular intake of beta blockers or calcium channel blockers
* Patients with any known hypersensitivity or contraindication to dexmedetomidine,
* Patients with significant neurological, psychiatric, or neuromuscular disorders.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2024-02-25 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-02 (Actual)

PRIMARY OUTCOMES:
Rate of successful intubations which was defined as both excellent and acceptable conditions. | 15 minutes
  * Excellent conditions: received a score of 1 for all the 5 factors.
  * Acceptable conditions: received a score of 2 for any of the 5 factors. Both excellent and acceptable conditions was defined as successful intubations. Poor conditions was defined as failed intubations.
  * Excellent conditions: received a score of 1 for all the 5 factors.
  * Acceptable conditions: received a score of 2 for any of the 5 factors. Both excellent and acceptable conditions was defined as successful intubations. Poor conditions was defined as failed intubations.

CONTACTS AND LOCATIONS:
Locations (1):
- Theodor Bilharz research institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No